CLINICAL TRIAL: NCT06781502
Title: Electronic Archive of Internal Medicine for the Treatment of Severe Organ Failure and Liver Transplantation-MITIGO
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: MITIGO
Record Dates: First submitted 2024-12-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-10

CONDITIONS: Organ Failure, Multiple; LIVER TRANSPLANTATION
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
ELECTRONIC ARCHIVE OF INTERNAL MEDICINE FOR THE TREATMENT OF SERIOUS ORGAN FAILURES AND LIVER TRANSPLANTATION

DETAILED DESCRIPTION:
This is an observational, spontaneous, monocentric study with structured data collection from the medical records of patients diagnosed with acute or chronic liver failure. The study will involve both retrospective and prospective data collection:

Retrospective data collection: Patients diagnosed between 01/01/2013 and the start date of the study.

Prospective data collection: Patients diagnosed after the start of the study until the end of the recruitment period (10 years).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute or chronic liver disease or LT
* Age ≥ 18 years
* Obtaining informed consent

Exclusion Criteria:

* no one

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients belonging to the U.O. will be enrolled. of the Liver Transplant Program of the IRCCS University Hospital of Bologna (Internal Medicine Unit for the treatment of serious organ failure, U.O. Hepatobiliary and Transplant Surgery, Program Abdominal surgery in end organ failure and in patients with organ transplant), in which a diagnosis of acute or chronic liver disease has been made or undergoing liver transplant, starting from 01/01/2013.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-10-21 (Actual); Primary Completion 2033-10 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Epidemiological classification of Acute or Chronic Liver Disease and Liver Transplant Candidates at the U.O. of Internal Medicine | 10 years
  This indicator will evaluate the main diagnostic states and substates of patients with acute or chronic liver disease and/or liver transplantation, followed at the U.O. of Internal Medicine for serious organ failure and the Liver Transplant Program of the IRCCS AOUBO.
Incidence of Complications in Chronic Liver Disease | 10 years
  This measure aims to assess the incidence of complications associated with chronic liver disease in patients followed at the U.O. of Internal Medicine and the Liver Transplant Program of the IRCCS AOUBO.
Hospitalization Rates | 10 years
  This section analyzes the hospitalization rates of patients with acute and chronic liver diseases, highlighting the frequency of hospital stays.
Number of Liver Transplantation Candidates Evaluated | 10 years
  This measure tracks the number of patients evaluated for liver transplantation at the U.O. of Internal Medicine and the Liver Transplant Program of the IRCCS AOUBO
Number of Liver Transplants Performed Annually | 10 years
  This measure tracks the number of liver transplants performed annually at the U.O. of Internal Medicine and the Liver Transplant Program of the IRCCS AOUBO.

SECONDARY OUTCOMES:
Description of Prescribed Treatments and Variations for Acute or Chronic Liver Disease and Liver Transplant Candidates at the U.O. of Internal Medicine | 10 years
  This measure aims to describe the prescribed treatments and any variations made for the entire population of patients with acute or chronic liver disease and/or liver transplantation, followed at the U.O. of Internal Medicine for serious organ failure and the Liver Transplant Program of the IRCCS AOUBO. Treatment data will be collected, including the specific therapies prescribed at diagnosis and during follow-up, as well as any modifications to the treatment plan based on patient response or clinical changes
Survival Rate Quantification | 10 years
  This measure aims to quantify survival rates for the entire population of patients with acute or chronic liver disease and/or liver transplantation, followed at the U.O. of Internal Medicine for serious organ failure and the Liver Transplant Program of the IRCCS AOUBO. Survival outcomes will be assessed starting from diagnosis, with rates measured at 1, 3, 5, and 10 years post-diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Vitale, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS - Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy